CLINICAL TRIAL: NCT04079803
Title: A Phase 2b, Randomized, Double-blind, Placebo-controlled, Multiple Dose, Biomarker and Safety Study of PTI-125 in Mild-to-moderate Alzheimer's Disease Patients
Brief Title: PTI-125 for Mild-to-moderate Alzheimer's Disease Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Cassava Sciences, Inc. (Industry)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PTI-125-02; R44AG060878 (NIH)
Record Dates: First submitted 2019-08-26; First posted 2019-09-06 (Actual); Results first posted 2021-06-01 (Actual); Last update posted 2021-09-29 (Actual); Status verified 2021-09

CONDITIONS: Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — Simufilam; Tablets

STUDY DESIGN:
Intervention Model Description: Approximately sixty (60) patients will be enrolled into the study and randomized to one of three cohorts. Cohorts will receive placebo or PTI-125 at 50 or 100 mg b.i.d. (n=20 per group)
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The sponsor, participant, care provider, investigator including sub-investigators and outcomes assessors will be blinded to throughout the study which includes using an Integrated Web Response System (IWRS) and electronic data capture (EDC) to ensure blinding during the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Placebo Cohort (Placebo Comparator): Subjects administered placebo oral tablets twice daily (BID)
  Interventions: Drug: Placebo oral tablet
- Simufilam (PTI-125) 100 mg tablets Cohort (Experimental): Subjects administered simufilam (PTI-125) 100 mg oral tablets twice daily (BID)
  Interventions: Drug: Simufilam 50 mg oral tablet
- Simufilam (PTI-125) 50 mg tablets Cohort (Experimental): Subjects administered simufilam (PTI-125) 50 mg oral tablets twice daily (BID)
  Interventions: Drug: Simufilam 100 mg tablet

INTERVENTIONS:
Drug: Placebo oral tablet — Oral placebo tablet
  Arms: Placebo Cohort
Drug: Simufilam 100 mg tablet — Simufilam 100 mg oral tablet
  Other Names: PTI-125
  Arms: Simufilam (PTI-125) 50 mg tablets Cohort
Drug: Simufilam 50 mg oral tablet — Simufilam 50 mg oral tablet
  Other Names: PTI-125
  Arms: Simufilam (PTI-125) 100 mg tablets Cohort

SUMMARY:
This is a Phase 2b, Randomized, Double-blind, Placebo-controlled, multiple dose study of PTI-125 in mild-to-moderate Alzheimer's disease patients.

DETAILED DESCRIPTION:
This is a Phase 2b, Randomized, Double-blind, Placebo-controlled, multiple dose study of PTI-125 in mild-to-moderate Alzheimer's disease patients. A total of sixty (60) patients will be enrolled in the study. Patients will receive Placebo, 50 mg or 100 mg b.i.d. of PTI-125. The objective of this study are to investigate the safety, and biomarkers of PTI-125 following 28-day repeat oral administration.

ELIGIBILITY:
Inclusion Criteria:

* Ages >= 50 and <= 85 years
* Informed consent form (ICF) signed by the subject or legally acceptable representative.
* Clinical diagnosis of dementia due to possible or probable Alzheimer's disease
* Mini-Mental State Examination score >= 16 and <= 26 at screening
* If female, postmenopausal for at least 1 year
* Patient living at home, senior residential setting, or an institutional setting without the need for continuous (i.e. 24-h) nursing care
* General health status acceptable for participation in the study
* Fluency (oral and written) in English or Spanish
* If receiving memantine, rivastigmine, galantamine or an AChEI, receiving a stable dose for at least 3 months. If receiving donepezil, any dose lower than 23 mg once daily.
* The patient is a non-smoker for at least 3 years.
* The patient or legal representative must agree to comply with the drawing of blood samples and with a lumbar puncture and the drawing of cerebrospinal fluid samples.
* The patient has a ratio of total tau/Aβ42 in cerebrospinal fluid >= 0.28.
* Patient has a caregiver or legal representative responsible for administering the drug and recording the time.

Exclusion Criteria:

* Exposure to an experimental drug, experimental biologic or experimental medical device within the longer of 5 half-lives or 3 months before screening
* Enrollment in the previous PTI-125 trial
* A medical condition that would interfere with a lumbar puncture
* Residence in a skilled nursing facility and requiring 24 h care.
* Clinically significant laboratory test results
* Clinically significant untreated hypothyroidism
* Insufficiently controlled diabetes mellitus
* Renal insufficiency (serum creatinine > ULN)
* Malignant tumor within 3 years before screening (except squamous and basal cell carcinoma or cervical carcinoma in situ or localized prostate cancer or localized stage 1 bladder cancer)
* History of ischemic colitis or ischemic enterocolitis
* Unstable medical condition that is clinically significant in the judgment of the investigator
* Alanine transaminase (ALT) or aspartate transaminase (AST) > ULN or total bilirubin > ULN.
* History of myocardial infarction or unstable angina within 6 months before screening
* History of more than 1 myocardial infarction within 5 years before screening
* Clinically significant cardiac arrhythmia (including atrial fibrillation), cardiomyopathy, or cardiac conduction defect (patients with a pacemaker are acceptable)
* Symptomatic hypotension, or uncontrolled hypertension
* Clinically significant abnormality on screening electrocardiogram (ECG), including but not necessarily limited to a confirmed corrected QT interval value >= 450 msec for males or >= 470 msec for females.
* Stroke within 18 months before screening, or history of a stroke concomitant with onset of dementia
* History of brain tumor or other clinically significant space-occupying lesion on CT or MRI
* Head trauma with clinically significant loss of consciousness within 12 months before screening or concurrent with the onset of dementia
* Onset of dementia secondary to cardiac arrest, surgery with general anesthesia, or resuscitation
* Specific degenerative Central Nervous System disease diagnosis other than Alzheimer's disease (eg, Huntington's disease, Creutzfeld-Jacob disease, Down's syndrome, Frontotemporal Dementia, Parkinson's disease)
* Wernicke's encephalopathy
* Active acute or chronic Central Nervous System infection
* Donepezil 23 mg quaque die currently or within 3 months prior to randomization
* Discontinued AChEI < 30 days prior to randomization
* Antipsychotics; low doses are allowed only if the subject has received a stable dose for at least 3 months before randomization
* Tricyclic antidepressants and monoamine oxidase inhibitors
* Anxiolytics or sedative-hypnotics, including barbiturates (unless given in low doses for benign tremor); low doses of benzodiazepines and zolpidem are allowed
* Immunosuppressants, including systemic corticosteroids, if taken in clinically immunosuppressive doses (Steroid use for allergy or other inflammation is permitted.)
* Antiepileptic medications if taken for control of seizures
* Chronic intake of opioid-containing analgesics
* Sedating H1 antihistamines
* Nicotine therapy (all dosage forms including a patch), varenicline (Chantix), or similar therapeutic agent within 30 days before screening
* Clinically significant illness within 30 days of enrollment
* History of significant neurological, hepatic, renal, endocrine, cardiovascular, gastrointestinal, pulmonary, or metabolic disease
* Positive serum hepatitis B surface antigen (HBsAg) or positive hepatitis C virus HCV antibody test at screening
* Positive HIV test at screening
* Positive urine drug test at screening
* Loss of a significant volume of blood (> 450 mL) within 4 weeks prior to the study
* Suicidality on C-SSRS at screening

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2019-09-09 (Actual); Primary Completion 2020-03-31 (Actual); Study Completion 2020-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lindsay Burns, PhD, Study Director — Cassava Sciences, Inc.
Locations (9):
- United States (9):
  - Cognitive Clinical Trials, Gilbert, Arizona
  - Cognitive Clinical Trials, Surprise, Arizona
  - Optimus U, Miami, Florida
  - IMIC, Inc., Palmetto Bay, Florida
  - Cognitive Clinical Trials, Bellevue, Nebraska
  - Cognitive Clinical Trials, Omaha, Nebraska
  - Advanced Memory Research Institute, Toms River, New Jersey
  - Centex Studies, Inc., Houston, Texas
  - Centex Studies, Inc., McAllen, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sever S. Role of actin cytoskeleton in podocytes. Pediatr Nephrol. 2021 Sep;36(9):2607-2614. doi: 10.1007/s00467-020-04812-z. Epub 2020 Nov 13. PMID 33188449
- See also: Altered filamin A enables amyloid beta-induced tau hyperphosphorylation and neuroinflammation in Alzheimer's disease — http://nnjournal.net/article/view/2313

RESULTS

PARTICIPANT FLOW:
Groups:
- Simufilam (PTI-125), 100 mg Tablets Cohort: Subjects administered simufilam 100 mg oral tablets twice daily (BID)
- Simufilam (PTI-125), 50 mg Tablets Cohort: Subjects administered simufilam 50 mg oral tablets twice daily (BID)
Period: Overall Study
Arm/Group | Placebo Cohort | Simufilam (PTI-125), 100 mg Tablets Cohort | Simufilam (PTI-125), 50 mg Tablets Cohort
Started | 22 | 21 | 21
Completed | 22 | 21 | 20
Not Completed | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Placebo Cohort: Subjects administered matching placebo tablets twice daily for 28 days.
- Simufilam (PTI-125), 100 mg Tablets Cohort: Subjects administered 100 mg simufilam tablets twice daily for 28 days.
- Simufilam (PTI-125), 50 mg Tablets Cohort: Subjects administered 50 mg simufilam tablets twice daily for 28 days.
- Total: Total of all reporting groups
Arm/Group | Placebo Cohort | Simufilam (PTI-125), 100 mg Tablets Cohort | Simufilam (PTI-125), 50 mg Tablets Cohort | Total
Number analyzed (Participants) | 22 | 21 | 21 | 64
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 4 | 9 | 6 | 19
  >=65 years | 18 | 12 | 15 | 45
Age, Continuous [Mean (Standard Deviation); unit: years] | 71.3 (6.68) | 69.3 (5.47) | 67.1 (8.76) | 69.2 (6.97)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 12 | 12 | 35
  Male | 11 | 9 | 9 | 29
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 9 | 11 | 11 | 31
  Not Hispanic or Latino | 13 | 10 | 10 | 33
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 2 | 2 | 4 | 8
  White | 19 | 19 | 17 | 55
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
CSF total tau/Aβ42 ratio [Mean (Standard Deviation); unit: ratio] | 1.20 (0.55) | 1.08 (0.50) | 1.17 (0.58) | 1.15 (0.54)
Mini-Mental State Exam (MMSE) [Mean (Standard Deviation); unit: units on a scale] — The MMSE is a is a widely used test of cognitive function among the elderly; it includes tests of orientation, attention, memory, language and visual-spatial skills. It is often used to stage Alzheimer's disease. The scale ranges from 0 to 30. No errors = 30.
  units on a scale | 23.1 (2.78) | 23.0 (2.66) | 22.7 (2.67) | 22.9 (2.70)
Taking cholinesterase inhibitor or memantine [Count of Participants; unit: Participants] | 8 | 7 | 5 | 20
Heterozygous APOE4 [Count of Participants; unit: Participants] | 12 | 14 | 9 | 35
Homozygous APOE4 [Count of Participants; unit: Participants] | 1 | 1 | 3 | 5
Paired Associates Learning total errors [Mean (Standard Deviation); unit: errors] — Boxes are displayed on the screen and are "opened" in a randomized order. One or more of them contains a pattern. The patterns are then displayed in the middle of the screen, one at a time and the participant must select the box in which the pattern was originally located. If the participant makes an error, the boxes are opened in sequence again to remind the participant of the locations of the patterns. The number of boxes increases progressively to a total of 8. Population: The least impaired patients (11 or fewer errors, representing a ceiling effect) and patients with 54 or more errors (very poor performance suggesting not understanding the task) were removed from the analysis. Also removed were the 3 patients with no detectable drug in plasma, 2 patients with ≥25% non-compliance by pill counts, one patient with no baseline test and one who did not understand instructions per rater notes.
  errors
    number analyzed (Participants) | 14 | 13 | 10 | 37
    (all) | 35.5 (19.65) | 31.0 (20.74) | 36.1 (18.76) | 34.2 (19.7)
Spatial Working Memory total errors [Mean (Standard Deviation); unit: errors] — A number of colored squares (boxes) are shown on the screen. By selecting the boxes and using a process of elimination, the subject should find one yellow 'token' in each of a number of boxes and use them to fill up an empty column on the right-hand side of the screen. The number of boxes is gradually increased to a total of 8 for the subjects to search. The colors and positions of the boxes are changed from trial to trial to discourage stereotyped search strategies. Population: Removed from analysis were the 3 patients with no detectable drug in plasma, 2 patients with ≥25% non-compliance by pill counts, one patient with no baseline test and one who did not understand instructions per rater notes
  errors
    number analyzed (Participants) | 22 | 18 | 17 | 57
    (all) | 19.0 (7.49) | 22.1 (5.88) | 22.3 (6.64) | 21.1 (6.67)
CSF Aβ42 [Mean (Standard Deviation); unit: pg/mL] — Population: One subject is missing a CSF sample. Three others had no detectable simufilam in plasma and were excluded from analyses.
  pg/mL
    number analyzed (Participants) | 22 | 19 | 18 | 59
    (all) | 125 (152) | 117 (51.4) | 108 (54.8) | 111 (86.1)
CSF total tau [Mean (Standard Deviation); unit: pg/mL] — Population: One subject is missing a CSF sample. Three others had no detectable simufilam in plasma and were excluded from analyses.
  pg/mL
    number analyzed (Participants) | 22 | 19 | 18 | 59
    (all) | 104 (32) | 106 (27.9) | 101 (17.6) | 103.7 (25.8)
CSF P-tau181 [Mean (Standard Deviation); unit: pg/mL] — Population: One subject is missing a CSF sample. Three others had no detectable simufilam in plasma and were excluded from analyses.
  pg/mL
    number analyzed (Participants) | 22 | 19 | 18 | 59
    (all) | 28.5 (0.73) | 29.7 (1.5) | 29.0 (1.0) | 29.1 (1.3)
CSF neurogranin [Mean (Standard Deviation); unit: pg/mL] — Population: One subject is missing a CSF sample. Three others had no detectable simufilam in plasma and were excluded from analyses.
  pg/mL
    number analyzed (Participants) | 22 | 19 | 18 | 59
    (all) | 1200 (365) | 1551 (751) | 1352 (614) | 1368 (577)
CSF Neurofilament Light Chain [Mean (Standard Deviation); unit: pg/mL] — Population: One subject is missing a CSF sample. Three others had no detectable simufilam in plasma and were excluded from analyses.
  pg/mL
    number analyzed (Participants) | 22 | 19 | 18 | 59
    (all) | 161 (42.8) | 219 (95.3) | 181 (64.4) | 187 (67.5)
CSF YKL-40 [Mean (Standard Deviation); unit: pg/mL] — Population: One subject is missing a CSF sample. Three others had no detectable simufilam in plasma and were excluded from analyses.
  pg/mL
    number analyzed (Participants) | 22 | 19 | 18 | 59
    (all) | 206 (29.5) | 203 (22.7) | 194 (26.0) | 201 (26.1)
CSF IL-6 [Mean (Standard Deviation); unit: pg/mL] — Population: One subject is missing a CSF sample. Three others had no detectable simufilam in plasma and were excluded from analyses.
  pg/mL
    number analyzed (Participants) | 22 | 19 | 18 | 59
    (all) | 32.5 (1.2) | 33.6 (1.8) | 33.6 (1.7) | 33.2 (1.6)
CSF sTREM2 [Mean (Standard Deviation); unit: pg/mL] — Population: One subject is missing a CSF sample. Three others had no detectable simufilam in plasma and were excluded from analyses.
  pg/mL
    number analyzed (Participants) | 22 | 19 | 18 | 59
    (all) | 878 (435) | 861 (421) | 882 (476) | 874 (444)
CSF HMGB1 [Mean (Standard Deviation); unit: pg/mL] — Population: One subject is missing a CSF sample. Three others had no detectable simufilam in plasma and were excluded from analyses.
  pg/mL
    number analyzed (Participants) | 22 | 19 | 18 | 59
    (all) | 424 (48.0) | 446 (67.3) | 454 (70.6) | 441 (62.0)
CSF/plasma albumin ratio [Mean (Standard Deviation); unit: ratio] — Population: One subject is missing a CSF sample. Three others had no detectable simufilam in plasma and were excluded from analyses.
  ratio
    number analyzed (Participants) | 22 | 19 | 18 | 59
    (all) | 0.24 (0.03) | 0.25 (0.08) | 0.25 (0.05) | 0.25 (0.05)
CSF/plasma IgG ratio [Mean (Standard Deviation); unit: ratio] — Population: One subject is missing a CSF sample. Three others had no detectable simufilam in plasma and were excluded from analyses.
  ratio
    number analyzed (Participants) | 22 | 19 | 18 | 59
    (all) | 0.200 (0.07) | 0.217 (0.11) | 0.227 (0.07) | 0.215 (0.08)
Lymphocyte filamin A - α7nAChR, Ratio to total filamin A [Mean (Standard Deviation); unit: ratio] — Population: One subject is missing a CSF sample. Three others had no detectable simufilam in plasma and were excluded from analyses.
  ratio
    number analyzed (Participants) | 22 | 19 | 18 | 59
    (all) | 0.59 (0.10) | 0.69 (0.11) | 0.66 (0.12) | 0.65 (0.11)
Lymphocyte filamin A - TLR4, Ratio to total filamin A [Mean (Standard Deviation); unit: ratio] — Population: One subject is missing a CSF sample. Three others had no detectable simufilam in plasma and were excluded from analyses.
  ratio
    number analyzed (Participants) | 22 | 19 | 18 | 59
    (all) | 0.55 (0.10) | 0.60 (0.07) | 0.58 (0.11) | 0.58 (0.09)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in CSF Abeta42
Description: Change from Baseline (screening sample) to Day 28 in cerebrospinal fluid levels of Amyloid beta42
Time Frame: Screening to Day 28
Population: As noted in the Participant Flow, one subject in the 50 mg arm did not complete the study. One additional subject in the 50 mg arm was missing a Day 28 CSF sample. This primary analysis includes one 50 mg subject who showed no detectable simufilam in plasma at return visits (their exclusion was not prespecified in the Statistical Analysis Plan).
Measure: Mean (Standard Deviation); unit: pg/mL
Groups:
- Placebo Cohort: Placebo tablets BID for 28 days
- Simufilam (PTI-125), 100 mg Tablets Cohort: simufilam 100 mg tablets BID for 28 days
- Simufilam (PTI-125), 50 mg Tablets Cohort: simufilam 50 mg tablets BID for 28 days
Arm/Group | Placebo Cohort | Simufilam (PTI-125), 100 mg Tablets Cohort | Simufilam (PTI-125), 50 mg Tablets Cohort
Number analyzed (Participants) | 22 | 21 | 19
pg/mL | 4.8 (30.9) | 12.5 (11.9) | 16.2 (21.1)
Statistical Analysis 1: Comparison: Placebo Cohort vs Simufilam (PTI-125), 100 mg Tablets Cohort; This primary analysis includes two 100 mg subjects who showed no detectable simufilam in plasma at return visits (their exclusion was not prespecified in the Statistical Analysis Plan); Test type: Superiority; p = 0.087, ANCOVA — P value adjusted for multiplicity of 6 co-primary endpoints (p<0.008 required for significance); General Linear Model for the analysis of covariance (ANCOVA) with a two-sided 95% confidence interval and baseline measurement as the covariate; In a secondary analysis removing two subjects with no detectable simufilam in plasma, P=0.0088 and CFB was 13.4. In percent change from baseline with these two subjects removed, P=0.004
Statistical Analysis 2: Comparison: Placebo Cohort vs Simufilam (PTI-125), 50 mg Tablets Cohort; This primary analysis includes one 50 mg subject who showed no detectable simufilam in plasma at return visits (their exclusion was not prespecified in the Statistical Analysis Plan); Test type: Superiority; p = 0.01, ANCOVA — P value adjusted for multiplicity of 6 co-primary endpoints (p<0.008 required for significance); [statistical method as in outcome 1, analysis 1]; In a secondary analysis removing one subject with no detectable simufilam in plasma, P=0.0006 and CFB was 16.9. In percent change from baseline with this subject removed, P=0.0004

2. Primary Outcome: Change From Baseline in CSF Total Tau.
Description: Change from Baseline (screening sample) to Day 28 in cerebrospinal fluid total tau.
Time Frame: Screening to Day 28
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: pg/mL
Groups:
- Placebo Cohort: Placebo oral tablets administered twice daily (BID)
- Simufilam (PTI-125) 100 mg Tablets Cohort: Simufilam (PTI-125) 100 mg oral tablets administered twice daily (BID)
- Simufilam (PTI-125) 50 mg Tablets Cohort: SImufilam (PTI-125) 50 mg oral tablets administered twice daily (BID)
Arm/Group | Placebo Cohort | Simufilam (PTI-125) 100 mg Tablets Cohort | Simufilam (PTI-125) 50 mg Tablets Cohort
Number analyzed (Participants) | 22 | 21 | 19
pg/mL | -3.2 (14.8) | -18.7 (10.4) | -14.6 (9.6)
Statistical Analysis 1: Comparison: Placebo Cohort vs Simufilam (PTI-125) 100 mg Tablets Cohort; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.0001, ANCOVA — P value adjusted for multiplicity of 6 co-primary endpoints (p<0.008 required for significance); [statistical method as in outcome 1, analysis 1]; In a secondary analysis removing two subjects with no detectable simufilam in plasma, P<0.0001 and CFB was -19.8
Statistical Analysis 2: Comparison: Placebo Cohort vs Simufilam (PTI-125) 50 mg Tablets Cohort; [analysis description as in outcome 1, analysis 2]; Test type: Superiority; p = 0.0012, ANCOVA — P value adjusted for multiplicity of 6 co-primary endpoints (p<0.008 required for significance); [statistical method as in outcome 1, analysis 1]; In a secondary analysis removing one subject with no detectable simufilam in plasma, P=0.001 and CFB was -14.9

3. Primary Outcome: Change From Baseline in CSF P-tau181
Description: Change from Baseline (screening) to Day 28 in cerebrospinal fluid P-tau181
Time Frame: Screening to Day 28
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Placebo Cohort | Simufilam (PTI-125), 100 mg Tablets Cohort | Simufilam (PTI-125), 50 mg Tablets Cohort
Number analyzed (Participants) | 22 | 21 | 19
pg/mL | -0.63 (1.8) | -3.1 (1.7) | -2.4 (1.6)
Statistical Analysis 1: Comparison: Placebo Cohort vs Simufilam (PTI-125), 100 mg Tablets Cohort; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.005, ANCOVA — P value adjusted for multiplicity of 6 co-primary endpoints (p<0.008 required for significance); [statistical method as in outcome 1, analysis 1]; In a secondary analysis removing two subjects with no detectable simufilam in plasma, P=0.003 and CFB was -3.2
Statistical Analysis 2: Comparison: Placebo Cohort vs Simufilam (PTI-125), 50 mg Tablets Cohort; [analysis description as in outcome 1, analysis 2]; Test type: Superiority; p = 0.002, ANCOVA — P value adjusted for multiplicity of 6 co-primary endpoints (p<0.008 required for significance); [statistical method as in outcome 1, analysis 1]; In a secondary analysis removing one subject with no detectable simufilam in plasma, P=0.003 and CFB was -2.5

4. Primary Outcome: Change From Baseline in CSF Neurogranin
Description: Change from Baseline (screening) to Day 28 in cerebrospinal fluid neurogranin
Time Frame: Screening to Day 28
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Placebo Cohort | Simufilam (PTI-125), 100 mg Tablets Cohort | Simufilam (PTI-125), 50 mg Tablets Cohort
Number analyzed (Participants) | 22 | 21 | 19
pg/mL | -50.5 (434) | -648 (491) | -527 (361)
Statistical Analysis 1: Comparison: Placebo Cohort vs Simufilam (PTI-125), 100 mg Tablets Cohort; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.0002, ANCOVA — P value adjusted for multiplicity of 6 co-primary endpoints (p<0.008 required for significance); [statistical method as in outcome 1, analysis 1]; In a secondary analysis removing two subjects with no detectable simufilam in plasma, P=0.0002 and CFB was -681
Statistical Analysis 2: Comparison: Placebo Cohort vs Simufilam (PTI-125), 50 mg Tablets Cohort; [analysis description as in outcome 1, analysis 2]; Test type: Superiority; p = 0.0005, ANCOVA — P value adjusted for multiplicity of 6 co-primary endpoints (p<0.008 required for significance); [statistical method as in outcome 1, analysis 1]; In a secondary analysis removing one subject with no detectable simufilam in plasma, P=0.0005 and CFB was -527

5. Primary Outcome: Change From Baseline in CSF Neurofilament Light Chain
Description: Change from Baseline (screening) to Day 28 in cerebrospinal fluid neurofilament light chain
Time Frame: Screening to Day 28
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Placebo Cohort | Simufilam (PTI-125), 100 mg Tablets Cohort | Simufilam (PTI-125), 50 mg Tablets Cohort
Number analyzed (Participants) | 22 | 21 | 19
pg/mL | -10.0 (45) | -76.3 (50.6) | -49.7 (35.5)
Statistical Analysis 1: Comparison: Placebo Cohort vs Simufilam (PTI-125), 100 mg Tablets Cohort; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.0003, ANCOVA — P value adjusted for multiplicity of 6 co-primary endpoints (p<0.008 required for significance); [statistical method as in outcome 1, analysis 1]; In a secondary analysis removing two subjects with no detectable simufilam in plasma, P=0.0002 and CFB was -78.5
Statistical Analysis 2: Comparison: Placebo Cohort vs Simufilam (PTI-125), 50 mg Tablets Cohort; [analysis description as in outcome 1, analysis 2]; Test type: Superiority; p = 0.0058, ANCOVA — P value adjusted for multiplicity of 6 co-primary endpoints (p<0.008 required for significance); [statistical method as in outcome 1, analysis 1]; In a secondary analysis removing one subject with no detectable simufilam in plasma, P=0.0008 and CFB was -51.0

6. Primary Outcome: Change From Baseline in CSF YKL-40
Description: Change from Baseline (screening) in cerebrospinal fluid YKL-40
Time Frame: Screening to Day 28
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Placebo Cohort | Simufilam (PTI-125), 100 mg Tablets Cohort | Simufilam (PTI-125), 50 mg Tablets Cohort
Number analyzed (Participants) | 22 | 21 | 19
pg/mL | -0.96 (24.2) | -22.3 (11.7) | -20.4 (17.4)
Statistical Analysis 1: Comparison: Placebo Cohort vs Simufilam (PTI-125), 100 mg Tablets Cohort; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.0001, ANCOVA — P value adjusted for multiplicity of 6 co-primary endpoints (p<0.008 required for significance); [statistical method as in outcome 1, analysis 1]; In a secondary analysis removing two subjects with no detectable simufilam in plasma, P=0.0001 and CFB was -23.7
Statistical Analysis 2: Comparison: Placebo Cohort vs Simufilam (PTI-125), 50 mg Tablets Cohort; [analysis description as in outcome 1, analysis 2]; Test type: Superiority; p = 0.0001, ANCOVA — P value adjusted for multiplicity of 6 co-primary endpoints (p<0.008 required for significance); [statistical method as in outcome 1, analysis 1]; In a secondary analysis removing one subject with no detectable simufilam in plasma, P=0.0002 and CFB was -20.9

7. Secondary Outcome: Paired Associates Learning Test
Description: Cognitive test assessing episodic memory. Boxes are displayed on the screen and are "opened" in a randomized order. One or more of them contains a pattern. The patterns are then displayed in the middle of the screen, one at a time and the participant must select the box in which the pattern was originally located. If the participant makes an error, the boxes are opened in sequence again to remind the participant of the locations of the patterns. The number of boxes increases progressively to a total of 8.
Time Frame: Day 1 to Day 28
Population: The least impaired patients (11 or fewer errors, representing a ceiling effect) and patients with 54 or more errors (very poor performance suggesting not understanding the task) were removed from the analysis. Also removed were the 3 patients with no detectable drug in plasma, 2 patients with ≥25% non-compliance by pill counts, one patient with no baseline test and one who did not understand instructions per rater notes.
Measure: Mean (Standard Deviation); unit: Change from Day 1 in total errors
Groups:
- Placebo Cohort: Placebo oral tablets administered twice daily (BID) for 28 days.
- Simufilam (PTI-125), 100 mg Tablets Cohort: Simufilam 100 mg oral tablets administered twice daily (BID) for 28 days.
- Simufilam (PTI-125), 50 mg Tablets Cohort: Simufilam 50 mg oral tablets administered twice daily (BID) for 28 days.
Arm/Group | Placebo Cohort | Simufilam (PTI-125), 100 mg Tablets Cohort | Simufilam (PTI-125), 50 mg Tablets Cohort
Number analyzed (Participants) | 14 | 13 | 10
Change from Day 1 in total errors | -1.5 (8.5) | -4.5 (17.7) | -5.7 (13.6)
Statistical Analysis 1: Comparison: Placebo Cohort vs Simufilam (PTI-125), 100 mg Tablets Cohort; This study was not powered for statistical significance on cognitive measures; Test type: Other; Effect size = 0.23 — Reported effect size vs. placebo was calculated with Hedge's g (for groups of 20 or fewer) but was identical when calculated by Cohen's d
Statistical Analysis 2: Comparison: Placebo Cohort vs Simufilam (PTI-125), 50 mg Tablets Cohort; This study was not powered for statistical significance on cognitive measures; Test type: Other; Effect size = 0.37 — [estimate comment as in outcome 7, analysis 1]

8. Secondary Outcome: Spatial Working Memory Test
Description: Cognitive assessment of spatial working memory: A number of colored squares (boxes) are shown on the screen. By selecting the boxes and using a process of elimination, the subject should find one yellow 'token' in each of a number of boxes and use them to fill up an empty column on the right-hand side of the screen. The number of boxes is gradually increased to a total of 8 for the subjects to search. The colors and positions of the boxes are changed from trial to trial to discourage stereotyped search strategies.
Time Frame: Day 1 to Day 28
Population: Removed from analysis were the 3 patients with no detectable drug in plasma, 2 patients with ≥25% non-compliance by pill counts, one patient with no baseline test and one who did not understand instructions per rater notes.
Measure: Mean (Standard Deviation); unit: Change from Day 1 in total errors
Groups:
- Simufilam (PTI-125), 100 mg Tablets Cohort: Simufilam, 100 mg oral tablets administered twice daily (BID)
- Simufilam (PTI-125), 50 mg Tablets Cohort: Simufilam, 50 mg oral tablets administered twice daily (BID)
Arm/Group | Placebo Cohort | Simufilam (PTI-125), 100 mg Tablets Cohort | Simufilam (PTI-125), 50 mg Tablets Cohort
Number analyzed (Participants) | 22 | 18 | 17
Change from Day 1 in total errors | -0.41 (7.54) | -2.31 (7.45) | -3.35 (4.86)
Statistical Analysis 1: Comparison: Placebo Cohort vs Simufilam (PTI-125), 100 mg Tablets Cohort; This study was not powered for statistical significance on cognitive measures; Test type: Other; Effect size = 0.46 — Reported effect size vs. placebo was calculated with Hedge's g (for groups of 20 or fewer) but was almost identical (0.45) when calculated by Cohen's d
Statistical Analysis 2: Comparison: Placebo Cohort vs Simufilam (PTI-125), 50 mg Tablets Cohort; This study was not powered for statistical significance on cognitive measures; Test type: Other; Effect size = 0.25 — [estimate comment as in outcome 7, analysis 1]

9. Secondary Outcome: CSF IL-6, sTREM2, HMGB1, Albumin, IgG
Description: Change from Baseline (screening sample) to Day 28 in secondary CSF biomarkers of neuroinflammation and blood-brain barrier integrity
Time Frame: Screening to Day 28
Population: Three subjects who had no detectable simufilam in plasma at return visits were removed from analyses (two in the 100 mg arm and one in the 50 mg arm). As noted in the Participant Flow, one subject in the 50 mg arm did not complete the study. One additional subject in the 50 mg arm was missing a Day 28 CSF sample.
Measure: Mean (Standard Deviation); unit: pg/mL; optical density for albumin & IgG
Arm/Group | Placebo Cohort | Simufilam (PTI-125), 100 mg Tablets Cohort | Simufilam (PTI-125), 50 mg Tablets Cohort
Number analyzed (Participants) | 22 | 19 | 18
pg/mL; optical density for albumin & IgG
  CSF IL-6 | -1.1 (2.0) | -3.7 (1.8) | -3.3 (1.9)
  CSF sTREM2 | -77.3 (510) | -426 (274) | -424 (386)
  CSF HMGB1 | 19.4 (172.3) | -143 (51.3) | -152 (50.1)
  CSF albumin | -240 (1620) | -2292 (1760) | -1245 (1735)
  CSF IgG | -574.8 (2518) | -2350 (2517) | -2444 (2097)
Statistical Analysis 1: Comparison: Placebo Cohort vs Simufilam (PTI-125), 100 mg Tablets Cohort; This analysis is for IL-6; Test type: Superiority; p = 0.0078, ANCOVA — Secondary CSF biomarkers were not adjusted for multiplicity; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Placebo Cohort vs Simufilam (PTI-125), 50 mg Tablets Cohort; This analysis is for IL-6; Test type: Superiority; p = 0.019, ANCOVA — Secondary CSF biomarkers were not adjusted for multiplicity; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Placebo Cohort vs Simufilam (PTI-125), 100 mg Tablets Cohort; This analysis is for sTREM2; Test type: Superiority; p = 0.0002, ANCOVA — Secondary CSF biomarkers were not adjusted for multiplicity; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: Placebo Cohort vs Simufilam (PTI-125), 50 mg Tablets Cohort; This analysis is for sTREM2; Test type: Superiority; p = 0.0007, ANCOVA — Secondary CSF biomarkers were not adjusted for multiplicity; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 5: Comparison: Placebo Cohort vs Simufilam (PTI-125), 100 mg Tablets Cohort; This analysis is for HMGB1; Test type: Superiority; p = 0.0001, ANCOVA — Secondary CSF biomarkers were not adjusted for multiplicity; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 6: Comparison: Placebo Cohort vs Simufilam (PTI-125), 50 mg Tablets Cohort; This analysis is for HMGB1; Test type: Superiority; p = 0.0001, ANCOVA — Secondary CSF biomarkers were not adjusted for multiplicity; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 7: Comparison: Placebo Cohort vs Simufilam (PTI-125), 100 mg Tablets Cohort; This analysis is for albumin; Test type: Superiority; p = 0.0001, ANCOVA — Secondary CSF biomarkers were not adjusted for multiplicity; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 8: Comparison: Placebo Cohort vs Simufilam (PTI-125), 50 mg Tablets Cohort; This analysis is for albumin; Test type: Superiority; p = 0.046, ANCOVA — Secondary CSF biomarkers were not adjusted for multiplicity; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 9: Comparison: Placebo Cohort vs Simufilam (PTI-125), 100 mg Tablets Cohort; This analysis is for Immunoglobulin G; Test type: Superiority; p = 0.012, ANCOVA — Secondary CSF biomarkers were not adjusted for multiplicity; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 10: Comparison: Placebo Cohort vs Simufilam (PTI-125), 50 mg Tablets Cohort; This analysis is for Immunoglobulin G; Test type: Superiority; p = 0.014, ANCOVA — Secondary CSF biomarkers were not adjusted for multiplicity; [statistical method as in outcome 1, analysis 1]

10. Other Pre Specified Outcome: Target Engagement Assays: Change From Baseline in Filamin A (FLNA) Linkages to alpha7 Nicotinic Acetylcholine Receptor (alpha7nAChR) and Toll-like Receptor 4 (TLR4) in Subject Lymphocytes
Description: FLNA linkages to these two receptors were assessed by densitometric quantitation of immunoblot bands of each receptor (detected by a specific antibody) in anti-FLNA precipitates. The measure is noted as a ratio to total FLNA.
Time Frame: Day 1 to Day 28
Population: Three subjects who had no detectable simufilam in plasma at any return visit were removed from analyses (two in the 100 mg arm and one in the 50 mg arm). As noted in the Participant Flow, one subject in the 50 mg arm did not complete the study. Two additional subjects in the 50 mg arm were missing Day 1 blood samples.
Measure: Mean (Standard Deviation); unit: ratio to total FLNA
Arm/Group | Placebo Cohort | Simufilam (PTI-125), 100 mg Tablets Cohort | Simufilam (PTI-125), 50 mg Tablets Cohort
Number analyzed (Participants) | 22 | 19 | 17
ratio to total FLNA
  FLNA - alpha7nAChR linkage | -0.07 (0.19) | -0.24 (0.16) | -0.23 (0.13)
  FLNA - TLR4 linkage | -0.05 (0.18) | -0.19 (0.14) | -0.19 (0.11)
Statistical Analysis 1: Comparison: Placebo Cohort vs Simufilam (PTI-125), 100 mg Tablets Cohort; Change from baseline in FLNA linkage to alpha7nAChR in subject lymphocytes. FLNA linkage to alpha7nAChR was expressed as the ratio of densitometric units of immunoblot bands of alpha7nAChR (probed with a specific antibody) to densitometric units of total FLNA; Test type: Superiority; p = 0.005, ANOVA — As secondary endpoints, lymphocyte biomarkers were not adjusted for multiplicity; ANOVA was used instead of ANCOVA due to the range in baseline values; it was deemed more appropriate to compare to each subject's own baseline value
Statistical Analysis 2: Comparison: Placebo Cohort vs Simufilam (PTI-125), 50 mg Tablets Cohort; Change from baseline in FLNA linkage to alpha7nAChR in subject lymphocytes. FLNA linkage to alpha7nAChR was expressed as ratios of densitometric units of immunoblot bands of alpha7nAChR (probed with a specific antibody) to densitometric units of total FLNA; Test type: Superiority; p = 0.009, ANOVA — As secondary endpoints, lymphocyte biomarkers were not adjusted for multiplicity; [statistical method as in outcome 10, analysis 1]
Statistical Analysis 3: Comparison: Placebo Cohort vs Simufilam (PTI-125), 100 mg Tablets Cohort; Change from baseline in FLNA linkage to TLR4 in subject lymphocytes. FLNA linkage to TLR4 was expressed as the ratio of densitometric units of immunoblot bands of TLR4 (probed with a specific antibody) to densitometric units of total FLNA; Test type: Superiority; p = 0.01, ANOVA — As secondary endpoints, lymphocyte biomarkers were not adjusted for multiplicity; [statistical method as in outcome 10, analysis 1]
Statistical Analysis 4: Comparison: Placebo Cohort vs Simufilam (PTI-125), 50 mg Tablets Cohort; [analysis description as in outcome 10, analysis 3]; Test type: Superiority; p = 0.01, ANOVA — As secondary endpoints, lymphocyte biomarkers were not adjusted for multiplicity; [statistical method as in outcome 10, analysis 1]

11. Other Pre Specified Outcome: Plasma P-tau181
Description: Percent change in plasma P-tau181
Time Frame: Day 1 to Day 28
Population: For plasma p-tau181 only: 4 subjects (1 in placebo, 2 in 50 mg and 1 in 100 mg arms) were removed because Coefficients of Variation (CVs) between duplicate measurements for either Day 1 or Day 28 samples were >15% on repeat assay (both Day 1 & Day 28 for a subject were repeated if CVs of either Day 1 or Day 28 were >11%). Two outliers were removed (1 in placebo [1.2 to 4.8 pg/ml] and 1 in 100 mg [2.1 to 5.1 pg/ml] arms) for increases >150% & > 2.5 pg/mL. Missing Day 1 blood samples: 2 in 50 mg.
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Placebo Cohort | Simufilam (PTI-125) 100 mg Tablets Cohort | Simufilam (PTI-125) 50 mg Tablets Cohort
Number analyzed (Participants) | 20 | 17 | 15
Percent change | 20.7 (49) | -16.5 (29) | -15.1 (36)
Statistical Analysis 1: Comparison: Placebo Cohort vs Simufilam (PTI-125) 100 mg Tablets Cohort; Test type: Superiority; p = 0.01, ANOVA; ANOVA followed by Dunnett's multiple comparisons test
Statistical Analysis 2: Comparison: Placebo Cohort vs Simufilam (PTI-125) 50 mg Tablets Cohort; Test type: Superiority; p = 0.02, ANOVA; ANOVA followed by Dunnett's multiple comparisons test
Statistical Analysis 3: Comparison: Placebo Cohort vs Simufilam (PTI-125) 100 mg Tablets Cohort vs Simufilam (PTI-125) 50 mg Tablets Cohort; Test type: Superiority; p = 0.009, ANOVA; This p value is for the main effect of treatment of the ANOVA

12. Other Pre Specified Outcome: Percent Change From Baseline in SavaDx, a Novel Plasma Biomarker
Description: SavaDx is a novel plasma biomarker
Time Frame: Day 1 to Day 28
Population: One subject in the 50 mg arm and two subjects in the 100 mg arm were omitted because these subjects showed no detectable plasma simufilam at any return visit. Two additional subjects in the 50 mg group were missing baseline plasma samples.
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Placebo Cohort | Simufilam (PTI-125), 100 mg Tablets Cohort | Simufilam (PTI-125), 50 mg Tablets Cohort
Number analyzed (Participants) | 22 | 19 | 17
Percent change | -3.2 (62) | -47.8 (19) | -44.1 (35)
Statistical Analysis 1: Comparison: Placebo Cohort vs Simufilam (PTI-125), 100 mg Tablets Cohort; Test type: Superiority; p = 0.003, ANOVA
Statistical Analysis 2: Comparison: Placebo Cohort vs Simufilam (PTI-125), 50 mg Tablets Cohort; Test type: Superiority; p = 0.016, ANOVA

ADVERSE EVENTS:
Time Frame: 28 days
Groups:
- Placebo Cohort: Subjects administered placebo tablets twice daily (BID) for 28 days.
- Simufilam (PTI-125), 100 mg Tablets Cohort: Subjects administered simufilam 100 mg tablets twice daily (BID) for 28 days.
- Simufilam (PTI-125), 50 mg Tablets Cohort: Subjects administered simufilam 50 mg tablets twice daily (BID) for 28 days.
Arm/Group | Placebo Cohort | Simufilam (PTI-125), 100 mg Tablets Cohort | Simufilam (PTI-125), 50 mg Tablets Cohort
All-Cause Mortality (participants affected / at risk) | 0/22 | 0/21 | 0/21
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/21 | 0/21
Other Adverse Events (participants affected / at risk) | 12/22 | 9/21 | 4/21
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo Cohort (N=22) | Simufilam (PTI-125), 100 mg Tablets Cohort (N=21) | Simufilam (PTI-125), 50 mg Tablets Cohort (N=21)
Headache (Nervous system disorders) | 3 (3) | 2 (2) | 1 (1)
Fatigue (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0)
Any adverse event (General disorders) | 12 (20) | 9 (15) | 4 (9)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (3):
  • Study Protocol (2019-06-28): https://cdn.clinicaltrials.gov/large-docs/03/NCT04079803/Prot_000.pdf
  • Statistical Analysis Plan (2020-02-12): https://cdn.clinicaltrials.gov/large-docs/03/NCT04079803/SAP_003.pdf
  • Informed Consent Form (2019-07-10): https://cdn.clinicaltrials.gov/large-docs/03/NCT04079803/ICF_002.pdf